CLINICAL TRIAL: NCT02912052
Title: Peri-operative Chemotherapy VS Postoperative Chemotherapy for the Treatment of Colon Cancer With Resectable Liver Metastasis: a Prospective Randomized Clinical Trial
Brief Title: Perioperative Chemotherapy VS Postoperative Chemotherapy for the Treatment of Colon Cancer With Resectable Liver Metastasis
Acronym: PEPCORLI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYM20160908
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Colon Cancer
Keywords: Perioperative Chemotherapy; Postoperative Chemotherapy; Colon Cancer; Resectable Liver Metastasis
MeSH Terms: conditions — Colonic Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peri-operative chemotherapy (Experimental): Patients receive 2 cycles of chemotherapy before surgery,and contniue to receive another 4 cycles of chemotherapy 21-28 days later after surgery.
  Interventions: Drug: Peri-operative chemotherapy
- postoperative chemotherapy (Active Comparator): Patients receive 6 cycles of chemotherapy 21-28 days later after surgery.
  Interventions: Drug: postoperative chemotherapy

INTERVENTIONS:
Drug: Peri-operative chemotherapy — Patients receive 2 cycles of chemotherapy before surgery,and contniue to receive another 4 cycles of chemotherapy 21-28 days later after surgery.The chemotherapy regime is XELOX(oxaliplatin130mg/m2 ivd d1 + Capecitabine1000mg/m2 po bid d1-14, 21d/cycle)
  Other Names: XELOX
  Arms: Peri-operative chemotherapy
Drug: postoperative chemotherapy — Patients receive 6 cycles of chemotherapy 21-28 days later after surgery.The chemotherapy regime is XELOX(oxaliplatin130mg/m2 ivd d1 + Capecitabine1000mg/m2 po bid d1-14, 21d/cycle)
  Other Names: XELOX
  Arms: postoperative chemotherapy

SUMMARY:
A prospective Randomized Clinical Trial to investigate the Effect ofPeri-operative Chemotherapy VS Postoperative Chemotherapy for the Treatment of Colon Cancer With Resectable Liver Metastasis

DETAILED DESCRIPTION:
Colon cancer (colorectal cancer CRC) is one of the most common malignant tumor of digestive tract, has become the global incidence of third malignant tumors, including colorectal cancer proportion increased year by year. With the way of life of residents in our country, the adjustment of diet and aging progress, the incidence of colorectal cancer is rising the trend, and most patients have been found in advanced disease. Tumor metastasis is an important factor affecting the prognosis of colon cancer, liver metastasis, especially, including simultaneous liver metastases and delayed liver metastasis from colon cancer, about 20% to 34% will appear at the same time of liver metastasis, about 40-50% of CRC patients died of liver metastasis at present, multi disciplinary team treatment to surgical treatment of the absolute dominance of the more and more attention, and benefit, but the optimum sequence of chemotherapy and surgery, is still unclear. The preoperative chemotherapy Potential advantages include: early treatment of micrometastasis; assessment of tumor response to chemotherapy (with prognostic value, contribute to the development of postoperative treatment plan); for those patients with early progression can avoid local treatment. Preoperative treatment of the potential disadvantages include: missed the surgery opportunity window period ", probably because in early stage of tumor progress, may also be because chemotherapy achieved complete remission and to determine the extent of resection surgery has become extremely difficult.2015 second edition of the NNCN guidelines that resectable metastatic disease initial resectable patients may be liver resection, adjuvant chemotherapy and postoperative; another alternative treatment mode is around perioperative chemotherapy (perioperative chemotherapy and postoperative chemotherapy). Therefore, gaps in the determination of the timing of chemotherapy is still the guide, worth exploring.

I center to carry out laparoscopic resection of colon cancer has been more than ten years, the accumulated number of cases more than 1000 cases, with rich experience of colon cancer. Comprehensive treatment including surgery, oncology, Radiology, pathology, Department of radiotherapy, a number of departments, the Department of endoscopy MDT team, and won the outstanding team of Chinese Medical Doctor Association in 2016 MDT honor.

This study used a prospective randomized method, evaluation of colon cancer with simultaneous resectable liver metastatic lesions and peri chemotherapy surgery after neoadjuvant chemotherapy of two therapeutic schemes for short-term and long-term effect, is expected to summarize the prospective data to support the operation and chemotherapy

ELIGIBILITY:
Inclusion Criteria:

(1) 18-80 years old, patients with synchronous liver metastatic colorectal cancer confirmed by pathology diagnosis(2) ASA score: I-III (3) MDT evaluation: primary tumor can be cut, liver metastases can get complete resection at R0 level. The adjacent Hepatic segments have enough blood flow to be shared and retain sufficient liver function, liver residual volume is larger than or equal to 50%; general condition of the patient is good enough, without extrahepatic unresectable metastasis, and can tolerate systemic chemotherapy. (4) there are evaluating lesions according to the RESIST 1 edition: at least the single path of the lesions can be accurately measured, and the maximum diameter of the conventional techniques (traditional physical examination, CT, X, MRI) ≥20mm CT≥10mm or spiral (5) within 3 weeks before entering the group , the laboratory test index and evaluation of the disease show good bone marrow, liver and kidney function reserve: 1) bone marrow function : Hb ≥ 90 g/L, neutrophil absolute value is more than 1.5 x 109/L, the platelet count was larger than 80 x 109/L; 2) renal function: serum creatinine < 1.5 x ULN or the creatinine clearance rate≥ 50 mL/min; 3) liver function: AST and ALT ≤2.5 *ULN(if the disease is caused by tumor, AST and ALT≤5 *ULN, hemobilirubin ≤2 *ULN. (6) signed the informed consent.

Exclusion Criteria:

(1) the pathological diagnosis is not adenocarcinoma or multiform pathological types. (2)with clinical symptoms requiring emergency surgery for treatment (complete obstruction, bleeding, intestinal perforation). (3) have received chemotherapy treatment or combined with other the anti-tumor treatment. (4) with serious basic diseases: heart disease, kidney failure, severe liver dysfunction or liver failure, coagulation dysfunction or oral dose of anticoagulant drugs, a baseline proteinuria (total urine protein >1g/d). (5) any other contraindications for the use of chemotherapy treatment (6) patients with pregnancy (7)with previous or existing central nervous system metastasis. (8) there have been cerebrovascular accident or stroke in the past 12 months (9) any other drugs may affect safety or surgical operation history (10) multiple primary colon cancer patients, or suffer from other malignant tumors, or have been systematic chemotherapy (11) with neurological or psychiatric disorders affecting cognitive ability (12)patients cannot accept the treatment because of the psychological, family or social reasons(13) patients with liver metastasis get complete remission after preoperative chemotherapy(14)patients with severe postoperative complications cannot do chemotherapy within the prescribed time (15)liver metastases cannot get hameochronous and R0 standard resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-10; Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Disease free survival，DFS | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

OTHER OUTCOMES:
recurrence-free survival | 5 years
local recurrence rate | 5 years
length of postoperative hospital stay | 30 days
early complication rate | 30 days
operative time | 1 day
number of lymph nodes retrieved | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Fumin Zhang, PHD, Study Director — Professor Ethics Committee of the First Affiliated Hospital, Nanjing Medical University, Jiangsu Province Hospital
Locations (1):
- Jiangsu province hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang ZM, Chen YY, Chen FF, Wang SY, Xiong B. Peri-operative chemotherapy for patients with resectable colorectal hepatic metastasis: A meta-analysis. Eur J Surg Oncol. 2015 Sep;41(9):1197-203. doi: 10.1016/j.ejso.2015.05.020. Epub 2015 Jun 11. PMID 26094113
- [Background] Bilchik AJ, Poston G, Adam R, Choti MA. Prognostic variables for resection of colorectal cancer hepatic metastases: an evolving paradigm. J Clin Oncol. 2008 Nov 20;26(33):5320-1. doi: 10.1200/JCO.2008.18.3152. Epub 2008 Oct 20. No abstract available. PMID 18936470
- [Background] Portier G, Elias D, Bouche O, Rougier P, Bosset JF, Saric J, Belghiti J, Piedbois P, Guimbaud R, Nordlinger B, Bugat R, Lazorthes F, Bedenne L. Multicenter randomized trial of adjuvant fluorouracil and folinic acid compared with surgery alone after resection of colorectal liver metastases: FFCD ACHBTH AURC 9002 trial. J Clin Oncol. 2006 Nov 1;24(31):4976-82. doi: 10.1200/JCO.2006.06.8353. PMID 17075115
- [Background] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Mauer M, Tanis E, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative FOLFOX4 chemotherapy and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC 40983): long-term results of a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1208-15. doi: 10.1016/S1470-2045(13)70447-9. Epub 2013 Oct 11. PMID 24120480
- [Background] Araujo R, Gonen M, Allen P, Blumgart L, DeMatteo R, Fong Y, Kemeny N, Jarnagin W, D'Angelica M. Comparison between perioperative and postoperative chemotherapy after potentially curative hepatic resection for metastatic colorectal cancer. Ann Surg Oncol. 2013 Dec;20(13):4312-21. doi: 10.1245/s10434-013-3162-8. Epub 2013 Jul 30. PMID 23897009
- [Background] Tamandl D, Gruenberger B, Herberger B, Kaczirek K, Gruenberger T. Surgery after neoadjuvant chemotherapy for colorectal liver metastases is safe and feasible in elderly patients. J Surg Oncol. 2009 Oct 1;100(5):364-71. doi: 10.1002/jso.21259. PMID 19235181
- [Background] Khoo E, O'Neill S, Brown E, Wigmore SJ, Harrison EM. Systematic review of systemic adjuvant, neoadjuvant and perioperative chemotherapy for resectable colorectal-liver metastases. HPB (Oxford). 2016 Jun;18(6):485-93. doi: 10.1016/j.hpb.2016.03.001. Epub 2016 Apr 20. PMID 27317952
- [Background] Schmoll HJ, Cartwright T, Tabernero J, Nowacki MP, Figer A, Maroun J, Price T, Lim R, Van Cutsem E, Park YS, McKendrick J, Topham C, Soler-Gonzalez G, de Braud F, Hill M, Sirzen F, Haller DG. Phase III trial of capecitabine plus oxaliplatin as adjuvant therapy for stage III colon cancer: a planned safety analysis in 1,864 patients. J Clin Oncol. 2007 Jan 1;25(1):102-9. doi: 10.1200/JCO.2006.08.1075. PMID 17194911
- [Background] Fong Y, Salo J. Surgical therapy of hepatic colorectal metastasis. Semin Oncol. 1999 Oct;26(5):514-23. PMID 10528899
- [Background] Muratore A, Zorzi D, Bouzari H, Amisano M, Massucco P, Sperti E, Capussotti L. Asymptomatic colorectal cancer with un-resectable liver metastases: immediate colorectal resection or up-front systemic chemotherapy? Ann Surg Oncol. 2007 Feb;14(2):766-70. doi: 10.1245/s10434-006-9146-1. Epub 2006 Nov 14. PMID 17103261
- [Background] Fong Y, Cohen AM, Fortner JG, Enker WE, Turnbull AD, Coit DG, Marrero AM, Prasad M, Blumgart LH, Brennan MF. Liver resection for colorectal metastases. J Clin Oncol. 1997 Mar;15(3):938-46. doi: 10.1200/JCO.1997.15.3.938. PMID 9060531